CLINICAL TRIAL: NCT00224146
Title: Multicenter Assessment of Transdermal Therapy in Overactive Bladder With Oxybutynin TDS (MATRIX)
Brief Title: Transdermal (TDS) Oxybutynin (Oxytrol(r)) in Overactive Bladder
Acronym: MATRIX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXY0402; MATRIX
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Overactive Bladder; Urinary Incontinence; Quality of Life
Keywords: Oxytrol(r); transdermal oxybutynin; overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

INTERVENTIONS:
Drug: oxybutynin transdermal delivery system (Oxytrol(r))

SUMMARY:
This study evaluates changes in health related quality of life outcomes in patients using Oxytrol(r)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with one or more symptom of overactive bladder, including urge urinary incontinence, urgency and/or frequency

Exclusion Criteria:

* Patients for whom Oxytrol(r) is contraindicated.
* Patients treated with Oxytrol(r) prior to participation in this study.
* Patients residing in long-term care facilities or nursing homes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2878 (Actual)
Dates: Start 2004-05; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Change in health-related quality of life

SECONDARY OUTCOMES:
Change in other outcomes such as:
depression
work productivity
participant satisfaction
effect of enhanced patient education on any of the above outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Naomi V. Dahl, PharmD, Study Director — Watson Laboratories, Inc.
Locations (10):
- United States (10):
  - Mobile, Alabama
  - Tucson, Arizona
  - Torrance, California
  - Rocky Hill, Connecticut
  - Valdosta, Georgia
  - Gretna, Louisiana
  - Bloomfield Hills, Michigan
  - Poughkeepsie, New York
  - Winston-Salem, North Carolina
  - Tomball, Texas

REFERENCES:
- [Result] Sand P, Zinner N, Newman D, Lucente V, Dmochowski R, Kelleher C, Dahl NV. Oxybutynin transdermal system improves the quality of life in adults with overactive bladder: a multicentre, community-based, randomized study. BJU Int. 2007 Apr;99(4):836-44. doi: 10.1111/j.1464-410X.2006.06658.x. Epub 2006 Dec 20. PMID 17187655
- [Result] Sand PK, Goldberg RP, Dmochowski RR, McIlwain M, Dahl NV. The impact of the overactive bladder syndrome on sexual function: a preliminary report from the Multicenter Assessment of Transdermal Therapy in Overactive Bladder with Oxybutynin trial. Am J Obstet Gynecol. 2006 Dec;195(6):1730-5. doi: 10.1016/j.ajog.2006.08.013. PMID 17132474
- [Result] Staskin DR, Rosenberg MT, Dahl NV, Polishuk PV, Zinner NR. Effects of oxybutynin transdermal system on health-related quality of life and safety in men with overactive bladder and prostate conditions. Int J Clin Pract. 2008 Jan;62(1):27-38. doi: 10.1111/j.1742-1241.2007.01625.x. Epub 2007 Nov 15. PMID 17983434